CLINICAL TRIAL: NCT03857152
Title: Can Contrast Enhanced Spectral Mammography (CESM) Reduce the Number of Benign Biopsies for Calcifications Without Negatively Impacting on Detection/Diagnosis of Clinically Significant Calcifications
Acronym: MICROENHANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RD17/91109
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient receiving CESM (Other): Patients will receive CESM in addition to normal standard treatment.
  Interventions: Diagnostic Test: Contrast enhanced spectral mammography (CESM)

INTERVENTIONS:
Diagnostic Test: Contrast enhanced spectral mammography (CESM) — Contrast enhanced spectral mammography (CESM) will be undertaken in addition to routine practice.
  CESM is a specialist mammography test that aims to 'highlight' areas of concern within the breast in more detail than a standard mammogram.
  The difference between CESM and a standard mammogram (x-ray of the breast) is the use of a special dye (called contrast medium) that is injected into the veins before the mammogram images are taken. The contrast enhanced images give more detailed information to the breast radiologists (expert doctors trained to analyse breast imaging).

SUMMARY:
Women who attend for their screening mammogram will be recalled if an abnormality is detected on the screening mammogram. Calcifications account for 20% of the women recalled to second stage screening. Currently there is no effective imaging tool to determine if the calcifications are cancer or not. Therefore, 90% of women will be subjected to a biopsy. 25-30% of the biopsies will show cancer. Contrast enhanced spectral mammography (CESM) is where contrast is given and then a mammogram performed. The theory is that high risk DCIS and invasive cancers have an increased blood supply and will therefore enhance more than benign lesions within the breast. If CESM can identify calcifications that are cancerous then we maybe able to reduce the number of women who have benign biopsies. This is patient focused as women would not require a biopsy and be able to be reassured at the same visit. This is also a cost-saving for the Trust by reducing unnecessary biopsies. This also supports the findings of the Marmot review by aiming to reduce harm by over-diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Recalled for second stage screening due to microcalcifications on the mammogram
2. Renal function is within normal limits
3. No known allergies to contrast
4. Able to give informed consent

Exclusion Criteria:

1. Known allergy to contrast
2. Renal impairment
3. Unable to provide informed consent
4. Having radioactive iodine treatment for hyperthyroidism

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-02-02 (Estimated); Study Completion 2021-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of benign biopsies | 3 years
  Total number of benign biopsies identified whilst undergoing CESM.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No